CLINICAL TRIAL: NCT07399132
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Part Study to Evaluate the Safety, Tolerability, and Immunogenicity of APL-10456-Vaccine in Healthy Volunteers
Brief Title: Phase 1 Study of APL-10456-Vaccine
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Apollo Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AP09CP01
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Rhinovirus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: in healthy volunteers age ≥18 years and ≤ 54 years Part B: in healthy volunteers ≥55 year (Experimental): Part A: Three (3) APL-10456-Vaccine dose levels which will be a sequential cohort single dose-escalation are planned, Part B will be a parallel group randomized controlled study to evaluate a two dose, prime and boost regimen of APL-10456-Vaccine in 3 dose levels
  Interventions: Drug: APL-10456-Vaccine
- Placebo (Placebo Comparator): Placebo is a comparator to Study Vaccine
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: APL-10456-Vaccine — 3 cohorts are planned for Part A and Part B
  Arms: Part A: in healthy volunteers age ≥18 years and ≤ 54 years Part B: in healthy volunteers ≥55 year
Other: Placebo — Placebo (a saline) is comparator to study vaccine
  Arms: Placebo

SUMMARY:
AP09CP01 is a Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Part Study which is conducted in Australia. The main purpose of this research study is to evaluate the safety, side effects, and immune response of APL-10456-Vaccine, a Rhinovirus (RV) Vaccine, when compared with a placebo in Younger and Older Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age Part A: Age ≥18 years and ≤54 years Part B: Age ≥55 years
* Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions of any type
* Acutely ill or febrile (temperature ≥38.0°C/100.4°F) 72 hours prior to or at the Day 1 visit
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, psychiatric or neurological disease/disorder within the past 3 months, or any acute minor illness (e.g. common cold, influenza, minor infection) within the past 1 month, determined by the PI (or delegate) to be clinically relevant
* Reported history of congenital or acquired immunodeficiency
* Dermatologic conditions that could affect local solicited AR assessments
* Coagulopathy or a bleeding disorder that is considered a contraindication to IM injection or phlebotomy
* Diagnosis of a malignancy within previous 5 years
* Has received systemic immunosuppressants for >14 days in total within 180 days prior to the Randomization Visit
* Has received or plans to receive any licensed or authorized vaccine, including COVID-19 vaccines, ≤28 days prior to the study injection (Day 1) or plans to receive a licensed or authorized vaccine within 28 days after the final study injection
* Has received systemic immunoglobulins, long-acting biological therapies that affect immune responses (eg, infliximab), or blood products within 90 days prior to the Randomization Visit or plans to receive them during the study
* Female participant with positive pregnancy test or Lactating females
* Has positive serology tests result (HIV, HCV and HBsAg) at screening visit
* Has positive drugs of abuse test results at screening visit
* Has participated in an interventional clinical study within 3 months prior to the Randomization Visit or plans to do so while participating in this study
* Has donated ≥450 mL of blood products within 28 days prior to the Randomization Visit or plans to donate blood products during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and reactogenicity of APL-10456-Vaccine in healthy volunteers (HVs) | Through Study Completion (Approx 365 days)
  Collecting AEs in Part A: HVs from 18 to 54 years of age, inclusive and Part B: HVs ≥ 55 years of age. Incidence, severity, relationship and outcome of Adverse Events (AE)

SECONDARY OUTCOMES:
To assess the immunogenicity of a single dose of APL-10456-Vaccine in Part A and B, and a prime/boost administration of APL-10456-Vaccine in Part B | Day 8 and Day 29 in Part A and approximately monthly visits up to Day 365 in Part B
  serotype-specific anti-APL-10456 antibody (IgG) titers and seroconversion rates in serum samples

IPD SHARING:
Plan to Share IPD: No